CLINICAL TRIAL: NCT05272904
Title: The QUILT Study: Quilting Sutures in Patients Undergoing Breast Cancer Surgery: a Stepped Wedge Cluster Randomized Trial Study
Brief Title: The QUILT Study: Quilting Sutures in Patients Undergoing Breast Cancer Surgery
Acronym: QUILT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Canisius-Wilhelmina Hospital (Other)
Collaborators: Rijnstate Hospital (Other); OLVG (Network); Martini Hospital Groningen (Other); Catharina Ziekenhuis Eindhoven (Other); St Jansdal Hospital (Other); Bravis Hospital (Other); Diakonessenhuis, Utrecht (Other); St. Antonius Hospital (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Principal Investigator, Lotte van Zeelst, Executive investigator, Canisius-Wilhelmina Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QUILT 2021-1
Record Dates: First submitted 2021-12-30; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Seroma
Keywords: Mastectomy; Breast cancer surgery; Quilting; Flap fixation; Seroma; Complications; Shoulder function; Pain; Cosmetic outcome; Health care consumption
MeSH Terms: conditions — Seroma; Pain

STUDY DESIGN:
Intervention Model Description: The QUILT study is a stepped wedge cluster randomized study.
Masking Description: Surgical technique is not blinded for surgeon and/or patients. An independent panel of four surgeons will blindly assess cosmetics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional closure method (Active Comparator): Following mastectomy, skin is closed using subcutaneous sutures followed by intracutaneous running suture. Depending on the surgeons discretion a vacuum closed suction drain was placed beneath the skin flaps.
  Interventions: Procedure: Conventional wound closure
- Quilting (Experimental): The implemented intervention is the quilting suture technique. The subcutaneous tissue is sutured to the pectoralis muscle placing multiple rows of running sutures. The suture starts at either end of the scar, running back and forth, creating rows of quilting stiches. The rows are placed transversely from the cranial to the caudal end of the wound with 2-3 cm between them, totalling some three to ﬁve rows for the cranial ﬂap. The caudal ﬂap is quilted with 2-3 rows in a caudal to cranial fashion. A subcutaneous suture followed by a intracutaneous running suture is used to close the skin. No wound drain is placed.
  Interventions: Procedure: Quilting

INTERVENTIONS:
Procedure: Quilting — Following mastectomy and/or axillary lymph node dissection, the subcutaneous tissue is sutured to the pectoralis muscle placing multiple rows of running sutures. The suture starts at either end of the scar, running back and forth, creating rows of quilting stiches. The rows are placed transversely from the cranial to the caudal end of the wound with 2-3 cm between them, totalling some three to ﬁve rows for the cranial ﬂap. The caudal ﬂap is quilted with 2-3 rows in a caudal to cranial fashion. A subcutaneous suture followed by a intracutaneous running suture is used to close the skin.
  Arms: Quilting
Procedure: Conventional wound closure — Following mastectomy, skin is closed using subcutaneous sutures followed by intracutaneous running suture. Depending on the surgeons discretion a vacuum closed suction drain was placed beneath the skin flaps.
  Arms: Conventional closure method

SUMMARY:
Seroma is the most common complication following breast cancer surgery, with reported incidence up to 90%. Seroma causes patient discomfort, is associated with surgical site infections (SSI), often requires treatment and increases healthcare consumption. The quilting technique, in which the skin flaps are sutured to the pectoralis muscle, leads to a significant reduction of seroma with a decrease in the number of aspirations and surgical site infections. Main objective of this randomized stepped wedge study is to assess the impact of large scale implementation of the quilting technique in patients undergoing mastectomy and/or axillary lymph node dissection. This will be one of the first multicentre prospective studies in which quilting without postoperative wound drain is compared with conventional wound closure. The hypothesis is that quilting is a simple and cost-effective technique to increase textbook outcome. Moreover, it is expected that patient comfort is enhanced by quilting.

DETAILED DESCRIPTION:
Seroma is the most common complication following breast cancer surgery, with reported incidence up to 90%. Seroma causes patient discomfort, is associated with surgical site infections (SSI), often requires treatment and increases healthcare consumption. The quilting technique, in which skin flaps are sutured to the pectoralis muscle, leads to a significant reduction of seroma with a decrease in the number of aspirations and surgical site infections. However, implementation is lagging due to unknown side effects, increase in operation time and cost effectiveness. Main objective of this study is to assess the impact of large scale implementation of the quilting suture technique in patients undergoing mastectomy and/or axillary lymph node dissection (ALND).

The QUILT study is a stepped wedge design study performed among nine teaching hospitals in the Netherlands. The study consists of nine steps, with each step one hospital will implement the quilting suture technique. Allocation of the order of implementation will be randomization-based. Primary outcome is 'textbook outcome', i.e.no wound complications, no re-admission, re-operation or unscheduled visit to the outpatient clinic and use of analgesics is not increased postoperative. A total of 113 patients is required based on a sample size calculation.

This will be one of the first multicentre prospective studies in which quilting without postoperative wound drain is compared with conventional wound closure. The hypothesis is that quilting is a simple technique to increase textbook outcome, without increasing health care consumption. Moreover, the expectation is that patient comfort is enhanced by quilting.

ELIGIBILITY:
Inclusion Criteria:

* all patients >18 years of age undergoing mastectomy and/or axillary lymph node dissection
* be irrespective of the nature of the primary tumour: prophylactic, risk reducing, benign, in situ carcinoma and invasive primary or recurrent carcinoma will be eligible, irrespective of preoperative systemic therapy.

Exclusion Criteria:

* patients who objected to participation (letter of objection)
* mentally incompetent patients or otherwise unable to complete a questionnaire
* immediate breast reconstruction
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Textbook outcome | 6 months
  'Textbook outcome' (TO), a combination of outcome parameters reflecting an ideal surgical outcome. Measured 6 months post-operative, the patients postoperative course must comply with the following to meet the definition of TO:
  * no wound complications
  * no re-admissions in relation to primary surgery
  * no re-operation in relation to primary surgery, re-excisions in case of involved margins allowed
  * no unscheduled visit to the outpatient clinic (depending on the centre one or two postoperative visits are usually scheduled)
  * postoperative use of analgesics (6 months) is not increased compared to pre-operative

SECONDARY OUTCOMES:
All palpation-detected seromas | 6 months
  Severity of complicaties are scored using the Clavien Dindo Classification of Surgical complications (grade I-V).
Clinical significant seroma | 6 months
  All aspirated seroma. Severity of complicaties are scored using the Clavien Dindo Classification of Surgical complications (grade I-V).
Surgical site infections | 6 months
  Severity of complicaties are scored using the Clavien Dindo Classification of Surgical complications (grade I-V).
Bleeding complications | 6 months
  Severity of complicaties are scored using the Clavien Dindo Classification of Surgical complications (grade I-V).
Wound healing problems | 6 months
  Including skin flap necrosis, wound necrosis, wound dehiscence. Severity of complicaties are scored using the Clavien Dindo Classification of Surgical complications (grade I-V).
Duration of surgery | 360 minutes
  Duration of surgery in minutes.
Length of hospital stay | 6 months
  Length of hospital stay in days: distinguishing between outpatient and inpatient treatment.
Unscheduled visits to the outpatient clinic | 6 months
  Number of unscheduled visits to the outpatient clinic
Readmission to the hospital | 6 months
  Readmission to the hospital related to primary surgery
Reoperation | 6 months
  Reoperation related to primary surgery other than re-excision.
Shoulder function | 6 months
  Assessed using the Disability of the Arm, Shoulder and Hand (DASH) questionnaire. Higher scores mean a worse outcome.
Post-operative pain | 14 days
  Assessed using the visual analogue scale (VAS). Scale 1-10, higher scores mean a worse outcome.
Post-operative pain | 6 months
  Post-operative use of analgesics (paracetamol, NSAID's, opioids).
Cosmetic outcome assessed by an independent panel | 6 months
  an independent panel of four surgeons will blindly assess cosmetics by classifying standardised digital photographs one a 4-point Likert scale with the following categories: poor, fair, good and excellent. Photos are taken in two positions: the first in neutral position with both arms hanging next to the body and the second with both arms raised in 180gr (or as far as possible) elevation.
Patient reported satisfaction with breast | 6 months
  BreastQ questionnaire for mastectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the study are available from the first and senior author on reasonable request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Zeelst LJV, Plate JDJ, van Eekeren RRJP, Ten Wolde B, Kroeze EMA, Schalken EC, de Wilt JHW, Strobbe LJA. Quilt technique after mastectomy: stepped-wedge randomized cluster trial showing superior textbook outcome and reduced healthcare utilization. Br J Surg. 2025 Sep 2;112(9):znaf175. doi: 10.1093/bjs/znaf175. PMID 41026907